CLINICAL TRIAL: NCT03152955
Title: Efficacy and Safety of Multimodal Analgesia Used in Patients With Microvascular Decompression
Brief Title: Postoperative Analgesia in Patients With Microvascular Decompression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XiangyaHospital
Record Dates: First submitted 2017-05-04; First posted 2017-05-15 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2017-05

CONDITIONS: Trigeminal Neuralgia
Keywords: trigeminal neuralgia; nerve block
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Ketamine; Ondansetron; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Patients in Group A will receive scalp nerve block and patient-controlled analgesia which contains sufentanil and ondansetron.
  Interventions: Other: scalp nerve block; Drug: ondansetron; Drug: Sufentanil
- Group B (Experimental): In Group B, patient-controlled analgesia which contains sufentanil、ondansetron and ketamine will be applied.
  Interventions: Drug: Ketamine; Drug: ondansetron; Drug: Sufentanil
- Group C (Sham Comparator): In Group C, patient-controlled analgesia which contains sufentanil and ondansetron will be applied.
  Interventions: Drug: ondansetron; Drug: Sufentanil

INTERVENTIONS:
Drug: Ketamine — Ketamine will be applied in patient-controlled analgesia.
  Arms: Group B
Other: scalp nerve block — Scalp nerve block is performed for the blockade of the greater occipital, superficial cervical and lesser occipital nerves with 0.5% ropivacaine.
  Arms: Group A
Drug: ondansetron — Ondansetron(13ug/kg/h) is applied in patient-controlled analgesia.
Drug: Sufentanil — Sufentanil(0.02ug/kg/h) is applied in patient-controlled analgesia.

SUMMARY:
Perioperative pain is caused by a variety of harmful factors through multiple mechanisms, therefore, reasonable postoperative analgesia should be combined with drugs or measures of different mechanism , which is called multimodal analgesia. Multimodal analgesia could minimize side effects and achieve a better analgesic effect. Commonly used strategies of multimodal analgesia are oral analgesic drug, nerve block, patient controlled analgesia and so on. This study will observe the effect of multimodal analgesia on postoperative pain in patients with microvascular decompression and record side effects. Finally, it will provide technical support for the guidance of postoperative analgesia in patients of trigeminal neuralgia.

DETAILED DESCRIPTION:
The investigators will collect 90 cases which will be divided into 3 groups. Patients in Group A will receive scalp nerve block and patient-controlled analgesia which contains sufentanil and ondansetron. In Group B, patient-controlled analgesia which contains sufentanil, ondansetron and ketamine will be applied. In Group C, patient-controlled analgesia which contains sufentanil and ondansetron will be applied.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of trigeminal neuralgia plan to receive microvascular decompression
2. Age between 18 and 70, ASA classification between Ⅰ～Ⅲ
3. No severe liver and kidney disease, no blood coagulation dysfunction
4. No history of long-term opioid drugs usage, no drug addiction history
5. Patients are fully conscious, cooperation, understanding and voluntarily signed informed consent

Exclusion Criteria:

1. More than 20% of the total blood volume is lost in operation
2. Intracranial hematoma happens within 24 h after surgery
3. Secondary surgery patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-05-15 (Estimated); Study Completion 2018-05-15 (Estimated)

PRIMARY OUTCOMES:
visual analog scale score | 6 hour after operation

CONTACTS AND LOCATIONS:
Overall Officials: Xie Yongqiu, Study Director — Xiangya Hospital of Central South University in Changsha
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided